CLINICAL TRIAL: NCT05792605
Title: Comparison of Anterior Talofibular Ligament Morphology on the Affected and Unaffected Side by Ultrasound in Stroke Patients
Brief Title: ATFL Evaluation With Ultrasound in Stroke Patients
Acronym: ATFL
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Pınar Doğan, resident doctor, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 19
Record Dates: First submitted 2023-03-08; First posted 2023-03-31 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stroke Sequelae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ATFL thickness increases on the affected side of stroke patients and the homogeneous fibrillar structure is deteriorated.We aim to compare morphology of ATFL and Achilles tendon on the affected and unaffected sides using ultrasound in hemiplegic patients.

DETAILED DESCRIPTION:
Age, gender, BMI, time elapsed after the event (months), Brunstrom motor stages and Barthel Activities of Daily Living index of the patients will be recorded. Modified Ashworth Scale and Tardieu scale are used to determine the muscle tone in the gastrocnemius, soleus and tibialis posterior of the hemiplegic side.

ATFL and Achilles tendon will be evaluated using a 12 MHz linear probe of the Toshibo Aplio 500 USG device.ATFL and Achilles tendon signal will be evaluated with reference to contralateral features.

ATFL will be evaluated while the patient lying in the supine position with knee flexion and ankle slight plantarflexion and inversion.The probe will be placed anterolaterally between the lateral malleolus and the talus and a longitudinal image of the ATFL is obtained.

Achilles tendon will be evaluated with the patient lying in the prone position and the ankle at 90 degrees neutral.

ATFL and Achilles tendon signal will be evaluated and noted as homogeneous normal fibrillary structure or heterogeneous.All ultrasound measurements will be performed twice with the patients in the same position.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering cerebrovascular accident associated stroke for the first time with a cortical or subcortical unilateral ischemia or hemorrhage
* Patients over the age of 18

Exclusion Criteria:

* Patients who were medically unstable
* Patients who had Botulinum Toxin A injection into any muscle in the last 6 months
* Patients who had other systemic neuromuscular disease
* Patients who had a previous orthopedic or neuromuscular injury to the lower extremity
* Patients who had a skin lesion at the measurement site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who apply to the Physical Medicine and Rehabilitation Clinic of Gaziosmanpaşa Training and Research Hospital between 20.02.2023- 20.03.2023 and who had hemiplegia or hemiparesis after their first cerebrovascular accident (CVO) will be included.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Anterior talofibular ligament(ATFL) thickness | baseline
  ATFL will be evaluated using a 12 MHz linear probe of the Toshibo Aplio 500 USG device. The thickness in millimeters will be measured from the midpoint of the ligament on the affected and unaffected side. Thicknesses will be compared and whichever side is thicker will be considered as increased in thickness. Being thicker is worse, indicating degenerative process.
Visual assessment of anterior talofibular ligament(ATFL) signal | baseline
  ATFL signal on the affected and unaffected side will be compared with ultrasound. ATFL signal will be evaluated and noted as homogeneous normal fibrillary structure or heterogeneous. It is worse when the ligament and tendon lose their homogeneous fibrillar structure and gain a heterogeneous appearance.
Visual assessment of achilles tendon signal | baseline
  Achilles tendon signal on the affected and unaffected side will be compared with ultrasound. Achilles tendon signal will be evaluated and noted as homogeneous normal fibrillary structure or heterogeneous. It is worse when the ligament and tendon lose their homogeneous fibrillar structure and gain a heterogeneous appearance.

SECONDARY OUTCOMES:
Brunstrom motor recovery stage | baseline
  The Brunnstrom stage describes the sequence of motor development and reorganization of the brain after stroke which contains 3 items for the arm, the hand, and the leg. The stage ranges from 1 (maximum possible impairment) to 7 (no impairment). As the patient's condition improves, the stage increases.
Barthel Index | baseline
  The Barthel Index is an ordinal scale used to measure performance in activities of daily living. Ten variables describing activities of daily living and mobility are scored, a higher number being a reflection of greater ability to function independently. Total scores on the Barthel index may range from 0-100 points, with a maximum score of 100 points indicating better performance.

OTHER OUTCOMES:
Modified Ashworth Scale of gastrocnemius, soleus and tibialis posterior muscles | baseline
  The spasticity level of ankle will be measured by using Modified Ashworth Scale. It measures resistance during passive soft-tissue stretching. The total or maximum scores for the subscale is 4 and the minimum is 0 score. Higher scores indicates the higher the tone, lower score indicates less tone. 0 score indicates normal tone and no increase in tone, while 4 scores indicate affected part rigid in flexion or extension.
Tardieu scale of gastrocnemius, soleus and tibialis posterior muscles | baseline
  The spasticity level of ankle will also be measured by using Tardieu Scale. The purpose of this scale is to quantify spasticity by assessing the muscle's response to different stretch velocities and by determining the spasticity angle. The scale ranges from 0 to 5 points, where 0 is equal to absence of spasticity, 5 is equal to high degree of spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: ebru yilmaz yalcinkaya, Prof MD, Study Director — gaziosmanpasa training and research hospital
Locations (1):
- Gaziosmanpasa Training Ve Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildizgoren MT, Velioglu O, Demetgul O, Turhanoglu AD. Assessment of the Anterior Talofibular Ligament Thickness in Patients with Chronic Stroke: An Ultrasonographic Study. J Med Ultrasound. 2017 Jul-Sep;25(3):145-149. doi: 10.1016/j.jmu.2017.03.001. Epub 2017 Mar 23. PMID 30065479
- [Result] Kwon DR, Park GY. Differences in lateral ankle ligaments between affected and unaffected legs in children with spastic hemiplegic cerebral palsy. J Ultrasound Med. 2013 Feb;32(2):313-7. doi: 10.7863/jum.2013.32.2.313. PMID 23341388